CLINICAL TRIAL: NCT00692835
Title: Immediate Postoperative Course of Patients With Mini Video Assisted Total Thyroidectomy (miVAT) Versus Classic Total Thyroidectomy (cTT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Papavramidis Theodossis, Elected lecturer, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 333/12-5-2008
Record Dates: First submitted 2008-06-05; First posted 2008-06-06 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Goiter
Keywords: Goiter [C19.874.283]; Thyroid Neoplasms [C19.874.788]
MeSH Terms: conditions — Goiter

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Patients with mini Video Assisted Thyroidectomy (miVAT)
  Interventions: Procedure: Total Thyroidectomy (Mini Video Assisted Thyroidectomy)
- B (Active Comparator): Immediate postoperative course of patients with classic Thyroidectomy (cTT)
  Interventions: Procedure: Total Thyroidectomy (Classic Thyroidectomy)

INTERVENTIONS:
Procedure: Total Thyroidectomy (Mini Video Assisted Thyroidectomy) — Immediate postoperative course of patients with Thyroidectomy
  Arms: A
Procedure: Total Thyroidectomy (Classic Thyroidectomy) — Immediate postoperative course of patients with Thyroidectomy
  Arms: B

SUMMARY:
Protocol Synopsis

* Protocol title: Immediate postoperative course of patients with mini Video Assisted Thyroidectomy (miVAT) versus classic Thyroidectomy (cTT)
* Purpose: Comparison of the immediate postoperative course and complications of the patients using the two techniques
* Design: Prospective, single-center randomized study
* Patient Population: Male or female subjects 18 years of age or older with nodular goiter who are scheduled for total thyroidectomy (miVAT or T)
* No. of Subjects: 100 patients divided into two groups, estimated up to 1 year to enroll
* Duration of Treatment: During the operation
* Duration of Follow-up: Follow-up will be performed daily while hospitalized, and by phone till the 7th postoperative day
* Endpoints: To evaluate the safety and cost-effectiveness of each technique

DETAILED DESCRIPTION:
1.0 INTRODUCTION

Classic articles by Kocher, Halsted, Lahey, Crile and Riddell have provided surgeons with principles that have significantly reduced operative morbidity and mortality from thyroidectomy. Nowadays, surgery of the thyroid gland is considered safe with practically null mortality. Morbidity, although infrequent, is still a reason for concern. The complications directly attributed to total thyroidectomy are hypoparathyroidism, recurrent laryngeal nerve injury, hemorrhage, oesophageal perforation and trachea instability and perforation. Furthermore, other complications, related to the surgical technique, such as seroma or wound infection, may also occur.

Several techniques are employed in order to resect the suffering thyroid gland. Classic total thyroidectomy (cTT) is considered today, the golden standard of total thyroid resection for nodular goiter. One the other hand, new technologies and great experience of several surgeons gave recently birth to a new technique named mini Video Assisted Thyroidectomy (miVAT).

This protocol is designed to compare data in regards to cTT versus miVAT in the immediate postoperative period - hospitalization period.

2.0 OBJECTIVES

To compare the immediate postoperative course and complications of the patients using the two techniques (cTT and miVAT).

3.0 DESIGN AND STUDY POPULATION

The study is designed as a prospective randomized single center study. Any patient that is scheduled for a total thyroidectomy for nodular goiter with nodules less that 4cm will be offered participation in this study.

The study will be conducted until 100 patients are treated (50 in each group). It is estimated that it will take up to 1 year to enroll the patients and an additional one week to obtain the follow-up information

4.0 STUDY PROCEDURE

4.1 Pre-Surgery

Procedures preformed such as routine hospital examinations, antibiotic prophylactic treatment, anticoagulant treatment and diet will be according to the standard management protocol and will be recorded for the study. The following pre-surgery information will be recorded:

1. Demographic information including: Age, gender, ethnicity
2. Height, weight, BMI and ASA status
3. Behavioral history (Smoking, alcohol or drug use)
4. Preoperative labs (WBC, Ht, Hgb, SGOT, SGPT, LDH, Glc, Ure, Cre, K+, Na+, Ca2+,Mg2+, TP, ALB, fT3, fT4, TSH, PTH, PT, aPTT, INR)
5. Diagnosis including clinical observations and previous imaging results
6. FNA results (if any)
7. Medications
8. Current and past history of surgical and medical comorbidities
9. Vocal cord assessment by indirect laryngoscopy

4.2 Intra-operative

The surgeon will perform the preplanned operation. Each recurrent laryngeal nerve has to be identified and its activity has to be recorded with the help of an electrode. The following intraoperative variables will be recorded for all patients:

1. Surgery date
2. Left laryngeal nerve activity
3. Right laryngeal activity
4. Method of devascularization of right lobe
5. Method of devascularization of left lobe
6. Technical complications
7. Estimated blood loss
8. Duration of surgery
9. Difficulty of the operation (1=very difficult to 5=very easy)
10. Operation performed
11. Procedure related comments
12. Usage of drains (number and type)
13. Usage of haemostatic material

4.3 Pathology data form

The following pathology data will be recorded for all patients:

1. Post-operative diagnosis including pathology report
2. Weight of the gland
3. Dimensions of the gland

4.4 Postoperative follow-up

Follow-up evaluation will be performed every day while hospitalized. There will be a contact by phone - if the patient is not hospitalized- every day until the 7th postoperative day. The following information will be recorded for all patients while they are hospitalized:

1. Temperature (max for 24hour period)
2. Wound infection
3. Antibiotics
4. Oral analgesic
5. Parenteral narcotics
6. Tolerating liquid and solids
7. Average Pain score for patient resting and moving/day
8. Postoperative labs (WBC, Ht, Hgb, SGOT, SGPT, LDH, Glc, Ure, Cre, K+, Na+, Ca2+,Mg2+, TP, ALB, fT3, fT4, TSH, PTH, PT, aPTT, INR)
9. Date of hospital ready to be discharged and date discharged
10. Blood in the drains (if any)
11. Sign of hypoparathyroidism (Chvostek and Trousseau)
12. Vocal alterations by patient (voice completely altered=10 to voice not altered=1)
13. Vocal cord assessment by indirect laryngoscopy
14. Comments

5.0 COMPLICATIONS AND ADVERSE EVENTS

The investigator is required to notify the coordinator of any serious adverse events. The coordinator is also required to notify the Ethics Committee according to local regulations and requirements.

Serious Adverse Events include:

1. Death regardless of cause
2. Any-life-threatening event
3. Any hospitalization or prolongation of existing hospitalization
4. Any event that results in persistent or significant disability or incapacity to the patient.

6.0 STATISTICAL ANALYSIS

The objective of this study is to compare the T with the miVAT techniques concerning the immediate postoperative course of the patients in relation to complications during and post procedure.

Statistical analysis included description of these intraoperative and postoperative outcomes, and indication of patient characteristics associated with these outcomes.

In order to efficiently compare the two techniques random allocation of the patients within two groups (Group A=T and Group B=miVAT) was employed. All patient with even number were included in group A, while all patients with odd number were included in group B.

Since the study does not have pre-specified hypotheses all statistical analyses are exploratory and interpretation of results should be within this context.

7.0 DATA MONITORING PLAN

The coordinator will monitor all data accrual. Furthermore, the coordinator will review the progress of the clinical trial including safety data and ensure as possible that it is conducted, recorded and reported in accordance with the protocol, good clinical practice and the applicable regulatory requirements.

8.0 DATA CONFIDENTIALITY

Each patient ill be identified by his/her initials and a unique patient identification number. Source data will be stored with source documents. Only personnel responsible for collecting data and transcribing it into the case report forms will have access to the data. Records will remain on site in secure areas.

10.0 ETHICS

Prior to study institution review board (IRB) approval should be obtained. Any changes in the study protocol, informed consent forms, or investigator must be re-approved by the IRB. All patients enrolled in the study will provide their consent prior to entering the study. An informed consent form shall be signed and dated by the patient. The investigator will retain the forms as part of the study records.

This study will be executed in accordance with the Declaration of Helsinki, in agreement with the guidelines for conducting a clinical investigation in accordance with the principles of ICH GCP outlined in the E6 document. By signing the present protocol, participants in the study commit themselves to carry it out in accordance with local legal requirements.

11.0 INFORMED CONSENT

All eligible patients should have the capacity to provide an informed consent. The above described inclusion and exclusion criteria were designed to ensure the entry of the appropriate population of patients to this study and will be approved by the local IRB. Screening for these criteria will be conducted by the coordinator.

Eligible patients will be educated about the research proposal by a study investigator. To determine whether the patient has understood the issues, he/she will be asked to describe what the research entails and whether they have any questions. All questions will be addressed prior to enrollment. The patient can refuse participation in the study at any time.

A written informed consent form will be generated. For each patient, a case report form (CRF) will be completed, providing general medical information and history.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is over 18 years old
2. Patient scheduled for a non-emergency operation
3. Patient signs and dates a written informed consent form (ICF) and indicates an understanding of the study procedures

Exclusion Criteria:

1. Patient had a previous operation at the thyroid
2. Patient is participating in another clinical trial which may affect this study's outcomes
3. Patient in toxic condition (non euthyroid or hypothyroid )
4. Patient receiving anticoagulation treatment for other medical condition
5. Echographic evidence that the size at least one nodule is more than 4cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Postoperative course of patients | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- 3rd Department of Surgery, AHEPA University Hospital, Thessaloniki, Thessaloniki, Greece